CLINICAL TRIAL: NCT04788186
Title: BEta Blocker dEprescription Following Coronary Artery Bypass Graft sURGERy: Feasibility and Safety Pilot (BEEFBURGER Trial)
Brief Title: Beta Blocker De-prescription Following Coronary Artery Bypass Graft Surgery (BEEFBURGER Trial).
Acronym: BEEFBURGER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian VIGOUR Centre (Other)
Responsible Party: Principal Investigator, Jay Shavadia, Assistant Professor Cardiology, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UofS REB Bio#2639
Record Dates: First submitted 2021-02-19; First posted 2021-03-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease; Acute Myocardial Infarction; Coronary Artery Stenosis; ST Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction (NSTEMI)
Keywords: Beta Blocker drugs; coronary artery bypass graft; CABG; De-prescription
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: open-label, randomized pilot comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continue beta blocker therapy (No Intervention): Participants in this arm will continue their beta blocker therapy as per their usual clinical care
- De-prescribe beta blocker therapy (Experimental): Beta blocker therapy will be de-prescribed in this arm
  Interventions: Drug: De-prescribe beta blocker therapy

INTERVENTIONS:
Drug: De-prescribe beta blocker therapy — Participants will be de-prescribed for beta-blocker therapy.
  De-prescription will be performed as follows:
  * Half of pre-randomization dose for the first 3 days, then
  * Half of the above dose for the next 3 days, then discontinue
  Other Names: De-prescription
  Arms: De-prescribe beta blocker therapy

SUMMARY:
Beta-blockers have the greatest cardiovascular impact in patients with reduced heart function/heart failure and in reducing the peri-operative risk of atrial fibrillation. In patients without these high-risk features treated with coronary artery bypass graft (CABG) surgery, their continued long-term role is unclear.

DETAILED DESCRIPTION:
This is an open-label, non-inferiority, randomized comparison of beta-blocker continuation versus de-prescription at the 6-8 week follow-up following isolated and uncomplicated CABG at Royal University Hospital, Saskatoon.

Patients treated with isolated CABG (without valve repair/replacement) and discharged on a beta-blocker are eligible for recruitment if they have preserved systolic function (EF ≥45%) and no history of heart failure, atrial fibrillation/flutter, or an alternate compelling indication for beta-blocker therapy. After obtaining informed consent, eligible patients are randomly assigned at 6-8 weeks to one of the two treatment groups: continued beta-blocker therapy per their usual clinical care OR beta-blocker de-prescription as per the study protocol.

The primary objective of this study is to demonstrate recruitment feasibility for beta-blocker de-prescription 6-8 weeks following uncomplicated CABG. Exploratory outcomes include the composite of all-cause mortality, myocardial infarction, stroke, arrhythmia, and cardiovascular-related hospitalization (congestive heart failure, recurrent ischemia, arrhythmia [supraventricular including atrial fibrillation, and ventricular], syncope or need for pacemaker) over a 3-year follow up duration.

Other exploratory outcomes will include a change in the patient reported quality of life using the Short Form (SF) 36 and Euro Qol (EQ) 5D questionnaires and angina score using the Seattle Angina Questionnaire (SAQ).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years treated with index isolated CABG
* Able to consent to study
* On beta blocker therapy at the 6-8week visit
* LV systolic function (≥45% assessed within 6months of CABG date)

Exclusion Criteria:

* Prior heart failure with reduced ejection fraction (LVEF <45%)
* Pre- or peri-operative atrial fibrillation or flutter
* Peri-CABG stroke
* Unable to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality | 3 years
  All-cause death includes death resulting from both cardiovascular and non-cardiovascular causes.
Rate of spontaneous myocardial infarction | 3 Years
  All spontaneous (type 1) myocardial infarctions as per the Universal MI definition.
  Typical rise or fall of biochemical markers of myocardial necrosis to greater than twice the upper limit of normal (ULN). If markers were already elevated, and have not reached their peak then further elevation of a marker ≥50% of a previous value and >2X ULN is required. If biomarkers are stable or decreasing then a re-elevation of ≥ 20% and > 2X ULN is required.
  All also require meeting at least one of the following criteria:
  * Ischemic symptoms
  * Development of new pathological Q waves (distinct from index STEMI)
  * ECG changes of new ischemia or
  * Pathological evidence of MI
Rate of stroke | 3 Years
  On the basis of CT or MRI imaging or autopsy, stroke is classified as:
  * Ischemic stroke (including hemorrhagic transformation of ischemic stroke)
  * Hemorrhagic stroke (including intracerebral / intraparenchymal hemorrhage and subarachnoid hemorrhage)
  * Undetermined stroke (no imaging or autopsy available)
Rate of hospitalizations for heart failure | 3 Years
  Physician decision to treat heart failure with intravenous furosemide, if already on oral diuretics (for an alternate indication other than prior congestive heart failure (CHF*), a 50% dose increase) with New York Heart Association class III or IV symptoms plus at least one of the following:
  * Presence of pulmonary edema or pulmonary vascular congestion on chest radiograph thought to be due to heart failure
  * Rales reaching above the lower 1/3 of the lung fields thought to be due to heart failure or
  * Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) >18 mm Hg
    * Patients with a prior history of heart failure are not eligible for randomization.
Rate of cardiac arrhythmia | 3 Years
  Supraventricular (excluding atrial fibrillation)
  * Includes all forms of Supraventricular tachycardia (SVT) such as atrioventricular reentry tachycardia (AVRT), atrioventricular node reentry tachycardia (AVNRT), atrial tachycardia
  * Atrial fibrillation
  Any new finding of clinical atrial fibrillation lasting greater than 30 seconds plus at least one of the following:
  * ECG
  * Rhythm strip
  * If ECG document or Holter report is unavailable, clear physician diagnosis Ventricular Non-sustained or sustained ventricular tachycardia or ventricular fibrillation
Rate of syncope or need for permanent pacemaker | 3 Years
  Syncope suspicious for cardiac etiology requiring either hospitalization for ≥ 24 hours or needing an implantable monitoring device (such as loop recorder) or permanent pacemaker
Rate of recurrent myocardial ischemia | 3 Years
  Hospitalization or stay in the emergency department for ≥ 24 hours for myocardial ischemia or requiring unplanned revascularization

SECONDARY OUTCOMES:
Change in patient reported quality of life (QoL) using Euro Qol (EQ) 5D questionnaire | 3 years
  Change in scores will be used to describe differences in the quality of life between the two study arms (Continuation Vs De-prescription).
  The EQ-5D is a patient self-reported questionnaire scored from 0 (being the worst health state imaginable meaning worse outcome) to 100 (being the best health state imaginable meaning better outcome).
Change in patient reported quality of life using Short Form (SF) 36 questionnaire | 3 years
  Change in scores will be used to describe differences in the quality of life between the two study arms (Continuation Vs De-prescription).
  The SF-36 consists of eight scaled scores. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability (meaning worse outcome). The higher the score the less disability (meaning better outcome) i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in the patient reported angina score using the Seattle Angina Questionnaire (SAQ) | 3 years
  The Seattle Angina Questionnaire is the most sensitive, specific, and responsive health-related quality of life instrument for coronary artery disease. The SAQ is a self-administered, disease-specific measure for patients with CAD that is valid, reproducible, and sensitive to clinical change. Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Haissam Haddad, MD, FRCPC, Study Chair — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macle L, Cairns J, Leblanc K, Tsang T, Skanes A, Cox JL, Healey JS, Bell A, Pilote L, Andrade JG, Mitchell LB, Atzema C, Gladstone D, Sharma M, Verma S, Connolly S, Dorian P, Parkash R, Talajic M, Nattel S, Verma A; CCS Atrial Fibrillation Guidelines Committee. 2016 Focused Update of the Canadian Cardiovascular Society Guidelines for the Management of Atrial Fibrillation. Can J Cardiol. 2016 Oct;32(10):1170-1185. doi: 10.1016/j.cjca.2016.07.591. Epub 2016 Sep 6. PMID 27609430
- [Background] Gillis AM, Skanes AC; CCS Atrial Fibrillation Guidelines Committee. Canadian Cardiovascular Society atrial fibrillation guidelines 2010: implementing GRADE and achieving consensus. Can J Cardiol. 2011 Jan-Feb;27(1):27-30. doi: 10.1016/j.cjca.2010.11.003. PMID 21329859
- [Background] Thaper A, Kulik A. Rationale for administering beta-blocker therapy to patients undergoing coronary artery bypass surgery: a systematic review. Expert Opin Drug Saf. 2018 Aug;17(8):805-813. doi: 10.1080/14740338.2018.1504019. Epub 2018 Jul 27. PMID 30037300
- [Background] Vaishnava P, Eagle KA. Surgery. beta-Blockers--still a trusted ally or time for retirement? Nat Rev Cardiol. 2014 Sep;11(9):502-3. doi: 10.1038/nrcardio.2014.112. Epub 2014 Jul 29. PMID 25072904
- [Background] Rossello X, Pocock SJ, Julian DG. Long-Term Use of Cardiovascular Drugs: Challenges for Research and for Patient Care. J Am Coll Cardiol. 2015 Sep 15;66(11):1273-1285. doi: 10.1016/j.jacc.2015.07.018. PMID 26361160
- [Background] Park JJ, Kim SH, Kang SH, Yoon CH, Cho YS, Youn TJ, Chae IH, Choi DJ. Effect of beta-Blockers Beyond 3 Years After Acute Myocardial Infarction. J Am Heart Assoc. 2018 Mar 3;7(5):e007567. doi: 10.1161/JAHA.117.007567. PMID 29502101
- [Background] Puymirat E, Riant E, Aissaoui N, Soria A, Ducrocq G, Coste P, Cottin Y, Aupetit JF, Bonnefoy E, Blanchard D, Cattan S, Steg G, Schiele F, Ferrieres J, Juilliere Y, Simon T, Danchin N. beta blockers and mortality after myocardial infarction in patients without heart failure: multicentre prospective cohort study. BMJ. 2016 Sep 20;354:i4801. doi: 10.1136/bmj.i4801. PMID 27650822
- [Background] Dondo TB, Hall M, West RM, Jernberg T, Lindahl B, Bueno H, Danchin N, Deanfield JE, Hemingway H, Fox KAA, Timmis AD, Gale CP. beta-Blockers and Mortality After Acute Myocardial Infarction in Patients Without Heart Failure or Ventricular Dysfunction. J Am Coll Cardiol. 2017 Jun 6;69(22):2710-2720. doi: 10.1016/j.jacc.2017.03.578. PMID 28571635
- [Background] Shavadia JS, Holmes DN, Thomas L, Peterson ED, Granger CB, Roe MT, Wang TY. Comparative Effectiveness of beta-Blocker Use Beyond 3 Years After Myocardial Infarction and Long-Term Outcomes Among Elderly Patients. Circ Cardiovasc Qual Outcomes. 2019 Jul;12(7):e005103. doi: 10.1161/CIRCOUTCOMES.118.005103. Epub 2019 Jul 9. PMID 31284739
- [Background] Shavadia JS, Zheng Y, Green JB, Armstrong PW, Westerhout CM, McGuire DK, Cornel JH, Holman RR, Peterson ED. Associations between beta-blocker therapy and cardiovascular outcomes in patients with diabetes and established cardiovascular disease. Am Heart J. 2019 Dec;218:92-99. doi: 10.1016/j.ahj.2019.09.013. Epub 2019 Oct 20. PMID 31715435
- [Background] Tsujimoto T, Sugiyama T, Shapiro MF, Noda M, Kajio H. Risk of Cardiovascular Events in Patients With Diabetes Mellitus on beta-Blockers. Hypertension. 2017 Jul;70(1):103-110. doi: 10.1161/HYPERTENSIONAHA.117.09259. Epub 2017 May 30. PMID 28559400
- [Background] Bangalore S, Steg G, Deedwania P, Crowley K, Eagle KA, Goto S, Ohman EM, Cannon CP, Smith SC, Zeymer U, Hoffman EB, Messerli FH, Bhatt DL; REACH Registry Investigators. beta-Blocker use and clinical outcomes in stable outpatients with and without coronary artery disease. JAMA. 2012 Oct 3;308(13):1340-9. doi: 10.1001/jama.2012.12559. PMID 23032550
- [Background] da Graca B, Filardo G, Sass DM, Edgerton JR. Preoperative beta-Blockers for Isolated Coronary Artery Bypass Graft. Circ Cardiovasc Qual Outcomes. 2018 Dec;11(12):e005027. doi: 10.1161/CIRCOUTCOMES.118.005027. No abstract available. PMID 30557046
- [Background] Bjorklund E, Nielsen SJ, Hansson EC, Karlsson M, Wallinder A, Martinsson A, Tygesen H, Romlin BS, Malm CJ, Pivodic A, Jeppsson A. Secondary prevention medications after coronary artery bypass grafting and long-term survival: a population-based longitudinal study from the SWEDEHEART registry. Eur Heart J. 2020 May 1;41(17):1653-1661. doi: 10.1093/eurheartj/ehz714. PMID 31638654
- [Background] Kohsaka S, Miyata H, Motomura N, Imanaka K, Fukuda K, Kyo S, Takamoto S. Effects of Preoperative beta-Blocker Use on Clinical Outcomes after Coronary Artery Bypass Grafting: A Report from the Japanese Cardiovascular Surgery Database. Anesthesiology. 2016 Jan;124(1):45-55. doi: 10.1097/ALN.0000000000000901. PMID 26517856
- [Background] Brinkman W, Herbert MA, O'Brien S, Filardo G, Prince S, Dewey T, Magee M, Ryan W, Mack M. Preoperative beta-blocker use in coronary artery bypass grafting surgery: national database analysis. JAMA Intern Med. 2014 Aug;174(8):1320-7. doi: 10.1001/jamainternmed.2014.2356. PMID 24934977
- [Background] Booij HG, Damman K, Warnica JW, Rouleau JL, van Gilst WH, Westenbrink BD. beta-blocker Therapy is Not Associated with Reductions in Angina or Cardiovascular Events After Coronary Artery Bypass Graft Surgery: Insights from the IMAGINE Trial. Cardiovasc Drugs Ther. 2015 Jun;29(3):277-85. doi: 10.1007/s10557-015-6600-y. PMID 26071975
- [Background] Goldberger JJ, Bonow RO, Cuffe M, Liu L, Rosenberg Y, Shah PK, Smith SC Jr, Subacius H; OBTAIN Investigators. Effect of Beta-Blocker Dose on Survival After Acute Myocardial Infarction. J Am Coll Cardiol. 2015 Sep 29;66(13):1431-41. doi: 10.1016/j.jacc.2015.07.047. PMID 26403339
- [Background] Zhang H, Yuan X, Zhang H, Chen S, Zhao Y, Hua K, Rao C, Wang W, Sun H, Hu S, Zheng Z. Efficacy of Long-Term beta-Blocker Therapy for Secondary Prevention of Long-Term Outcomes After Coronary Artery Bypass Grafting Surgery. Circulation. 2015 Jun 23;131(25):2194-201. doi: 10.1161/CIRCULATIONAHA.114.014209. Epub 2015 Apr 23. PMID 25908770
- [Background] Allen JE, Knight S, McCubrey RO, Bair T, Muhlestein JB, Goldberger JJ, Anderson JL. beta-blocker dosage and outcomes after acute coronary syndrome. Am Heart J. 2017 Feb;184:26-36. doi: 10.1016/j.ahj.2016.10.012. Epub 2016 Oct 22. PMID 27892884